CLINICAL TRIAL: NCT04749433
Title: A Phase 1 Study to Assess the Safety and Tolerability of PET Imaging With [11C]CPPC [5-cyano-N-(4-(4-[11C]Methylpiperazin-1-yl)-2-(Piperidin-1-yl)Phenyl)Furan-2-carboxamide] Radioligand in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Study of [11C]CPPC to Assess the Safety and Tolerability in Patients With ALS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study stopped to enhance protocol and resume under different sponsor
Sponsor: Johns Hopkins University (Other)
Collaborators: Precision Molecular (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00263068
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Positron Emission Tomography
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: There will be two groups of participants in this study, healthy control participants and participants with a diagnosis of ALS. All patients will receive the same radiotracer and scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with diagnosis of ALS (Experimental): Participants with a diagnosis of ALS will receive a single dose of [11C]CPPC (370 megabecquerel (MBq) (X±1 mCi)) intravenously and subsequent positron emission tomography (PET) scan.
  Interventions: Drug: [11C]CPPC Injection
- Healthy Participants without a diagnosis of ALS (Experimental): Healthy participants (without a diagnosis of ALS) will receive a single dose of [11C]CPPC (370 megabecquerel (MBq) (X±1 mCi)) intravenously and subsequent positron emission tomography (PET) scan.
  Interventions: Drug: [11C]CPPC Injection

INTERVENTIONS:
Drug: [11C]CPPC Injection — A single dose of [11C]CPPC (370 megabecquerel (MBq) (X±1 mCi)) intravenously and subsequent positron emission tomography (PET) scan.
  Other Names: [5-cyano-N-(4-(4-[11C]methylpiperazin-1-yl)-2-(piperidin-1-yl)phenyl)furan-2-carboxamide]

SUMMARY:
The goal of this study is to evaluate the safety of using the [5-cyano-N-(4-(4-[11C]Methylpiperazin-1-yl)-2-(Piperidin-1-yl)Phenyl)Furan-2-carboxamide] ([11C]CPPC) radiotracer in positron emission tomography (PET) imaging of people with amyotrophic lateral sclerosis (ALS). The investigators are also interested to see whether use of this radiotracer reveals imaging differences between patients with ALS and healthy patients.

DETAILED DESCRIPTION:
This is a Phase 1 study of safety and tolerability of an investigational radiotracer drug called [5-cyano-N-(4-(4-[11C]Methylpiperazin-1-yl)-2-(Piperidin-1-yl)Phenyl)Furan-2-carboxamide] ([11C]CPPC). A radiotracer is a substance that chemically marks certain structures in the body. In this case, [11C]CPPC highlights structures expressing colony stimulating factor receptor (CSF1R), a receptor that is expressed on microglial cells. A safety and tolerability study is looking to see if there are any unanticipated, possibly harmful, effects of the use of the radiotracer in humans. However, ultimately, the investigators would like to know if this drug can be used to make better images of the brain for patients with amyotrophic lateral sclerosis (ALS), which could help doctors better understand the disease and help take care of patients with ALS. This study will use a radiotracer to look for a chemical receptor which ALS patients have more of in the brain. After receiving the radiotracer, participants' brains will be scanned with a positron emission tomography (PET) imaging machine.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, provide written informed consent, understand and provide written authorization for the use and disclosure of Protected Health Information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) Privacy Ruling] and comply with the study procedures.
2. Men and women at least 18 years old.
3. Women must have a negative serum pregnancy test and practice an acceptable method of contraception or be of non-childbearing potential (post-menopausal for at least 2 years or who have undergone hysterectomy, oophorectomy or surgical sterilization).
4. Geographic accessibility to the study center and the ability to travel to the clinic for study visits.
5. Presence of a willing and able caregiver.
6. Diagnosis of ALS based on examination by the site PI, meeting El Escorial criteria for possible, laboratory-supported probable, probable or definite ALS or be a person without a diagnosis of ALS disorder
7. Vital capacity ≥ 50% of predicted normal for age, height and gender measured in the seated position and the ability to lie supine for a period of 1 hour.
8. Agrees to the visit schedule as outlined in the informed consent.
9. Pre-study labs within normal range, or if abnormal, deemed not clinically significant by the site investigator.

Exclusion Criteria:

1. Weakness due to causes other than ALS.
2. Receipt of any investigational drug, device or biologic within 30 days of administration of study compound.
3. Use of anti-inflammatory medications, immunosuppressants, or benzodiazepines.
4. Any concomitant medical disease or condition limiting the safety to participate including, but not limited to:

   1. Coagulopathy
   2. Active infection
5. Any condition that the site PI feels may interfere with participation in the study
6. Inability to provide informed consent as determined by the site PI.
7. Known clinical evidence of frontotemporal dementia
8. Inadequate family or caregiver support as determined by the site PI.
9. Presence of any of the following conditions:

   1. Current drug abuse or alcoholism
   2. Unstable medical conditions
   3. Unstable psychiatric illness including psychosis and untreated major depression within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Safety of use of [11C]CPPC in patients with ALS as assessed by adverse events | Up to 10 days follow up after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by number of adverse events during and 10 days after the injection.
Safety of use of [11C]CPPC in patients with ALS as assessed by a change in neurological status | Baseline and 10 days after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by neurological physical exam to determine if there is a change in the findings from baseline.
Safety of use of [11C]CPPC in patients with ALS as assessed by a change in complete blood count (CBC) test | Baseline and 10 days after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by monitoring of the complete blood count (CBC) for a change from baseline that is outside of the normal range.
Safety of use of [11C]CPPC in patients with ALS as assessed by a change in complete metabolic panel (CMP) test | Baseline and 10 days after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by a change in the CMP from baseline that is outside of the normal range.

SECONDARY OUTCOMES:
Sensitivity of use of [11C]CPPC as assessed by a radiologist | 1 day
  Sensitivity of use of [11C]CPPC in PET neuroimaging to detect ALS will be determined by comparing the PET images from patients with ALS with those from healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Maragakis, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horti AG, Naik R, Foss CA, Minn I, Misheneva V, Du Y, Wang Y, Mathews WB, Wu Y, Hall A, LaCourse C, Ahn HH, Nam H, Lesniak WG, Valentine H, Pletnikova O, Troncoso JC, Smith MD, Calabresi PA, Savonenko AV, Dannals RF, Pletnikov MV, Pomper MG. PET imaging of microglia by targeting macrophage colony-stimulating factor 1 receptor (CSF1R). Proc Natl Acad Sci U S A. 2019 Jan 29;116(5):1686-1691. doi: 10.1073/pnas.1812155116. Epub 2019 Jan 11. PMID 30635412